CLINICAL TRIAL: NCT00102765
Title: A Multicenter, Randomized, Double-Blind, Parallel Group, 52-Week Comparison of Asthma Control and Measures of Airway Inflammation in Subjects of African Descent Receiving Fluticasone Propionate/Salmeterol 100/50mcg DISKUS® BID or Fluticasone Propionate 100mcg DISKUS® BID Alone
Brief Title: Study Of Asthma In Patients Of African Descent
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SFA103153
Record Dates: First submitted 2005-02-01; First posted 2005-02-02 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Asthma
Keywords: asthma exacerbation; asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: fluticasone propionate/salmeterol powder
Drug: fluticasone propionate powder
  Other Names: fluticasone propionate/salmeterol powder

SUMMARY:
This study will last up to 62 weeks. You will visit the clinic up to 17 times. Certain clinic visits will include physical examination, medical history review and lung function tests. The purpose of this study is to see if one asthma drug (fluticasone propionate/salmeterol) is better in reducing the number of asthma exacerbations compared with another drug (fluticasone propionate alone)

ELIGIBILITY:
Inclusion criteria:

* History of asthma for at least 6 months.
* Taking a low-dose of an inhaled corticosteroid for at least one month prior to the study (such as fluticasone propionate or budesonide).

Exclusion criteria:

* History of life-threatening asthma.
* Hospitalized for asthma within 3 months prior to the study.
* Current respiratory tract infection.
* Will not be able to attend clinic visits for the entire length of the study.
* Certain medical conditions that will make being in the study unsafe (such as congestive heart failure, uncontrolled hypertension, tuberculosis or certain drug allergies).

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 479 (Actual)
Dates: Start 2004-11; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Asthma exacerbation rate per patient per year

SECONDARY OUTCOMES:
Morning peak flow measurement, percent of asthma symptom-free days, percent of albuterol-free days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (64):
- United States (64):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Montgomery, Alabama
  - GSK Investigational Site, Muscle Shoals, Alabama
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Palmdale, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Stockton, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Hartford, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Martinez, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Flossmoor, Illinois
  - GSK Investigational Site, Lafayette, Louisiana
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Ypsilanti, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Picayune, Mississippi
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Verona, New Jersey
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, West Sayville, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Elizabeth City, North Carolina
  - GSK Investigational Site, High Point, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Sylvania, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Jenkintown, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Newport News, Virginia
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Bailey W, Castro M, Matz J, White M, Dransfield M, Yancey S, Ortega H. Asthma exacerbations in African Americans treated for 1 year with combination fluticasone propionate and salmeterol or fluticasone propionate alone. Curr Med Res Opin. 2008 Jun;24(6):1669-82. doi: 10.1185/03007990802119111. Epub 2008 May 6. PMID 18462564
- [Derived] Anderson WH, Koshy BT, Huang L, Mosteller M, Stinnett SW, Condreay LD, Ortega H. Genetic analysis of asthma exacerbations. Ann Allergy Asthma Immunol. 2013 Jun;110(6):416-422.e2. doi: 10.1016/j.anai.2013.04.002. PMID 23706709
- [Derived] Camargo CA Jr, Sutherland ER, Bailey W, Castro M, Yancey SW, Emmett AH, Stempel DA. Effect of increased body mass index on asthma risk, impairment and response to asthma controller therapy in African Americans. Curr Med Res Opin. 2010 Jul;26(7):1629-35. doi: 10.1185/03007995.2010.483113. PMID 20429821
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: SFA103153 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: SFA103153 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: SFA103153 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: SFA103153 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: SFA103153 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: SFA103153 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: SFA103153 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register